CLINICAL TRIAL: NCT03855436
Title: Identify Intermediate Coronary Lesions at High Risk of Progression-Study Design and Protocol of a Prospective Observational Study
Brief Title: Risk Factors of Intermediate Coronary Lesion Progression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: Intermediate Lesion
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Coronary Atheroscleroses; Coronary Angiography
Keywords: coronary intermediate lesions; quantitative flow reserve; serum biomarker; risk score
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary intermediate lesions generally refer to lumen narrowing with diameter stenosis% (DS%) between 50% and 70% on angiography. Prognosis varies significantly among patients with intermediate lesions, and some lesions progress rapidly leading to adverse cardiovascular events. Therefore, accurate risk stratification is important and will help clinicians identify patients at high risk of adverse events. The aim of study is to identify independent risk factors for major adverse cardiovascular events (MACE) among patients with intermediate lesions.

The study is a prospective, single-center, ongoing, observational study, which aims at enrolling approximately 1389 patients with intermediate coronary lesions. After enrollment, the following data are collected for each participant: baseline characteristics including demographics, clinical presentation, traditional risk factor, diagnosis and management; lesion characteristics assessed by coronary angiography; quantitative flow reserve; lab tests including blood chemistry, blood lipid, hemoglobin A1C, cardiac biomarker, BNP, et al. Patients are followed up at 2 year for primary outcome including death, myocardial infarction and repeat unplanned revascularization. A risk prediction score will be established and validated for major adverse cardiovascular disease at two-year follow-up.

DETAILED DESCRIPTION:
Study setting This ongoing study is conducted in Fuwai Hospital, one of the world's biggest cardiovascular center specializing in all kinds of cardiovascular diseases, particularly those complex, difficult, and severe cardiovascular diseases. More than 10000 angiographic procedures is performed each year in Fuwai Hospital.

Recruitment

From 2017 January 1st, all patients admitted to Fuwai Hospital receiving elective coronary angiography were screened for eligibility. Detailed inclusion and exclusion creteria are shown as follows:

Inclusion Criteria:

1. Receiving elective coronary angiography.
2. One or more lesions located in main coronary arteries with intermediate stenosis (defined as diameter stenosis of 50%-70%).
3. No lesions with significant stenosis (greater than 70%)

Exclusion criteria:

1. Unable to sign consent
2. Receiving percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
3. Planned PCI or CABG
4. Left ventricle ejection fraction % (LVEF%)<35% or cardiogenic shock
5. Other severe comorbidities with life expectancy <1 year

Data quality assurance Data are collected, submitted and stored online to the Informatics Center of Fuwai Hospital. Data are stored and protected managed according to national information security protection law. The following measures are adopted for data quality control. (1) Research staff will only be given access to a password-protected data-entry system after formal training. (2) A real-time, automated algorithm is used to check the logic, range, validity, consistency, completeness of data entered in the system. (3) Approximately 10% of online records are selected randomly and checked against the source documentation. (4) Data management team will check data quality regularly, and ask research staff to review and revise the missing, invalid and illogical data.

Missing data Several measures will be adopted to manage missing data: (1) "Required" fields are used for key variables during data entry. (2) We conducted pilot testing to identify variables with high rate of missing data, explore possible reasons and improve data collection. (3) Data management team will monitor data quality periodically and send queries to researchers to enter the missing data and check invalid data. (4) During statistical analysis phase, based on the type, pattern and amount of missing data, appropriated methods will be used to handle missing data.

Data collection Data are collected by trained experienced cardiologists and by using standardized definition in accordance with ACC/AHA Task Force on clinical Data Standards and NCDR-CathPCI registry Data Coder's Dictionary, including patient demographics, clinical presentation, medical history, risk factors, physical examination, laboratory results, clinical events, angiographic characteristics and procedural characteristics.

Quantitative flow ratio (QFR) QFR was calculated based on coronary angiography [9] and detailed algorithms for calculation have been described. In the first step, two angiographic images at the same cardiac phase, at least 25° apart, were selected and transferred to QFR system. A common anatomic landmark on two image frames was defined for system offset correction. The start and end point of the interrogated vessel was then defined, and lumen counters of the interrogated vessel were automatically delineated. In case of suboptimal image quality, manual correction was performed. In the next step, contrast-entry and contrast-exit frames for interrogated vessel were defined, followed by generation of QFR report.

Serum Biomarker Fasting blood samples were taken from cubital veins on the first day of admission, before and after coronary angiography procedure for biomarker and analysis. Serum and plasma are separated and stored in batches for analysis. Peripheral blood mononuclear cells are separated by centrifugation techniques and stored at -80°C. Full blood count, blood chemistry test including high sensitivity C-Reactive protein (hs-CRP), lipoprotein, creatinine, creatine kinase (CK), creatine kinase-MB (CK-MB), blood lipid, Na+, K+, glucose, N-terminal pro b-type natriuretic peptide (NT-proBNP), high-sensitive Troponin I (hsTnI) , troponin I (TnI), microalbumin urine test are performed as routine practice in Fuwai Hospital.

Follow-up All participants in this project are followed-up at 2 year by telephone call or e-mail. Vital status, adverse event, medication adherence, control of risk factors including smoking, BMI, blood pressure, blood lipid, blood glucose and physical activity are collected by trained staff using standardized form. If any adverse event is reported, medical records are reviewed carefully and adjudicated by independent clinicians.

Primary outcome measures The primary outcome was defined as major adverse cardiovascular events (MACE), which was defined as a composite of death, non-fatal myocardial infarction (MI) and unplanned repeat revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Receiving elective coronary angiography
* Written informed consent
* One or more lesions located in main coronary arteries with intermediate stenosis (defined as diameter stenosis of 50%-70%)
* No lesions with significant stenosis (greater than 70%)

Exclusion Criteria:

* Unable to sign consent
* Receiving percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
* Planned PCI or CABG
* Left ventricle ejection fraction % (LVEF%)<35% or cardiogenic shock
* Other severe comorbidities with life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suspected of CAD and underwent elective coronary angiogram. Patients have signed written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1389 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 2 years
  death, nonfatal myocardial infarction, repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD, PhD, Principal Investigator — National Center for Cardiovascular Diseases; Fuwai Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No